CLINICAL TRIAL: NCT03944616
Title: Effect of Artificially Sweetened Beverages on Diabetes Control in Adults With Type 2 Diabetes
Brief Title: Study Of Drinks With Artificial Sweeteners in People With Type 2 Diabetes
Acronym: SODAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Minnesota (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrew Odegaard, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20184756; 1R01DK117028-01A1 (NIH)
Record Dates: First submitted 2018-11-19; First posted 2019-05-09 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Diet beverages; diet; diabetes control; artificial sweeteners; continuous glucose monitor; gut microbiome; metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Artificially Sweetened Beverages; Water

STUDY DESIGN:
Intervention Model Description: This study is testing the effect of commercial diet beverage intake on diabetes control parameters in free-living adults with type 2 diabetes in a randomized, two arm parallel trial with a run-in period of 2-weeks and an active intervention period of 24-weeks. We will recruit 200 patients with type 2 diabetes who are usual consumers of commercial diet beverages and randomize them to receive and consume either: 1) A commercial diet beverage of choice (3 servings or 24 oz. daily); or 2) Unflavored bottled water of choice (sparkling or plain) (3 servings or 24 oz. daily).
Who Masked: Outcomes Assessor
Masking Description: All nursing staff/phlebotomist collecting physical samples, and the lab analyzing the samples will be masked to the trial arm the participant is in. The biostatistician performing the final analyses will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Beverage (Active Comparator): Participants will receive and consume three daily servings (24 ounces) of a non-caloric commercial diet beverage of their choice sweetened with FDA approved artificial sweeteners.
  Interventions: Behavioral: Diet Beverage
- Water (Experimental): Participants will receive and consume three daily servings (24 ounces) of plain bottled/canned water in place of their usual commercial diet beverage. The water will be unflavored, unsweetened, non-caloric, and may be plain or sparkling. Participants randomized to consume water will be instructed to avoid intake of diet beverages.
  Interventions: Behavioral: Water

INTERVENTIONS:
Behavioral: Diet Beverage — Participants will receive and consume three daily servings (24 ounces) of a non-caloric commercial diet beverage of their choice sweetened with FDA approved artificial sweeteners.
  Arms: Diet Beverage
Behavioral: Water — Participants will receive and consume three daily servings (24 ounces) of plain bottled/canned water in place of their usual commercial diet beverage. The water will be unflavored, unsweetened, non-caloric, and may be plain or sparkling. Participants randomized to consume water will be instructed to avoid intake of diet beverages.
  Arms: Water

SUMMARY:
Diet beverages sweetened with artificial sweeteners occupy a unique category in the food environment as they are a source of intensely sweet taste with no calories. Diet beverages are the single largest contributor to artificial sweetener intake in the U.S. diet, and people with diabetes are the highest consumers of diet beverages, tending to consume them as a replacement for dietary sources of sugar, especially in place of sugar-sweetened beverages. This behavior has been endorsed by dietetic and scientific organizations, and diet beverages are marketed as being synonymous with better health, suitable for weight loss, and thus advantageous for diabetes control. The underlying public health concern is that there are few data to support or refute the benefit or harm of habitual diet beverage consumption by people with diabetes; therefore randomized trials with relevant outcomes must be conducted because they would address many limitations of previous research and have major implications for dietary recommendations on diet beverage intake and primary and secondary prevention of chronic disease. To begin addressing this important scientific gap the investigators are testing the effect of diet beverage intake on diabetes control parameters in free-living adults with type 2 diabetes in a randomized, two arm parallel trial with a run-in period of 2-weeks and an active intervention period of 24-weeks. This study will recruit 200 patients with type 2 diabetes who are usual consumers of commercial diet beverages and randomize them to receive and consume either: 1) A commercial diet beverage of choice (3 servings or 24 oz. daily); or 2) Unflavored bottled water of choice (sparkling or plain) (3 servings or 24 oz. daily). The primary outcome will be a central measure of clinical diabetes control in glycated hemoglobin (HbA1c). The study will also measure the nature and magnitude of glycemic excursions via continuous glucose monitors, as well as clinical markers of cardiometabolic risk and kidney function. Lastly, investigators will measure plausible mechanisms whereby diet beverage intake may alter risk by assessing the effect of diet beverage intake on the functional composition of the gut microbiome via stool samples and comprehensive metabolomics, satiety hormones, as well as usual dietary intake, and upstream behavioral pathways which may inform dietary intake patterns.

ELIGIBILITY:
Inclusion criteria: We will include men, women and non-binary participants with T2D, age 35 years and older, able to provide informed consent, otherwise healthy, who meet the following criteria:

* Physician diagnosed type 2 diabetes ≥ 6 months prior to screening
* HbA1c 6.5-8.5% at participant screening
* Current treatment with lifestyle changes or stable diabetes-related medication levels for the past 3 months
* Willingness to provide consent to contact treating physician and physician agreement to refrain from changing diabetes-related medications during the trial (change defined as > 2 fold change in dose of any 1 hyperglycemic agent or addition or subtraction of an agent)
* No physician-directed medication change for 3 months if prescribed medication for lipids or blood pressure
* Usual consumers of diet beverages (≥ 3 servings/ week (24 oz.) and the willingness to maintain fidelity of the intervention, and participate in all aspects of the intervention
* Not actively looking to make major lifestyle alterations during the study period with stable weight for 2 months (within 3%).

Exclusion Criteria:

* Type 1 diabetes or suspected type 1 diabetes (lean with polyuria, polydipsia, and weight loss with little response to metformin)
* "Secondary" diabetes due to specific causes (e.g. monogenic syndromes, pancreatic surgery, and pancreatitis)
* Diabetic Ketoacidosis hospitalization within last 6 months
* Severe/major hypoglycemia in the last 3 months-severe/major hypoglycemia is defined as a hypoglycemic event in which patient requires assistance of another person to manage the episode
* Glucocorticoid use (prednisone 2.5 mg/d or more or its equivalent)
* History of intolerance or allergy to diet beverages or AS or phenylketonuria
* Any condition that is known to affect the validity of the glycemic measures (Hba1c)
* Major cardiovascular disease event or surgery within past 6 months
* Gastrointestinal disease
* Renal or liver disease
* Current treatment for cancer
* Those with major surgery planned or history of bariatric surgery
* Antibiotic treatment (> 6 days) within past 6 months
* Currently pregnant (via self-report) or planning to become pregnant during study period; <1 year postpartum and breast feeding
* Current participation in another interventional clinical trial
* Previous randomization in this study,
* Heavy alcohol consumption (on average >2 drinks/day for women and >3 drinks/day for men)
* Habitual consumer of SSB ≥ 1 serving / day (8 oz.)
* Does not drink diet beverages
* BMI < 20.0 kg/m2

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diet Beverage | Water
Started | 91 | 90
Completed | 91 | 88
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Beverage | Water | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.4) | 60.7 (10.1) | 60.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 44 | 43 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or Black | 4 | 2 | 6
  Hispanic/Latino(a) | 9 | 11 | 20
  White (non-Hispanic) | 68 | 67 | 135
  Other | 10 | 10 | 20
Region of Enrollment [Number; unit: participants] — States (California) and (Minnesota)
  participants
    United States | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Glycated hemoglobin
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: Participants analyzed at each time point equals: baseline (all those randomized to arm), 12 weeks (reflects those who were not able to participate in visit with blood draw to to Covid-19 restrictions and dropouts), and 24 weeks (all ASB participants provided data, 87 water participants (2 dropouts/lost to follow up and 1 with sample not able to be analyzed)
Measure: Mean (Standard Deviation); unit: Hba1c(%)
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
Hba1c(%)
  Time 0 | 7.19 (1.10) | 7.20 (0.69)
  12 weeks: number analyzed (Participants) | 86 | 84
  12 weeks | 7.13 (1.02) | 7.43 (1.02)
  24 weeks: number analyzed (Participants) | 91 | 87
  24 weeks | 7.14 (1.19) | 7.44 (1.04)

2. Secondary Outcome: Time In Range
Description: Time in range is collected by a masked Continuous Glucose Monitor (CGM), which measures individual glucose levels every 15 minutes for two weeks via a sensor placed on the participants upper arm (underside). Time in Range is defined as the % of time each day with a glucose measure between 70-180 mg/dl. The range of CGM data for inclusion in this study will be 5 to 14 days, consistent with manufacturer's recommendations.
Time Frame: All 14 day periods: Run-in (2-weeks, usual-baseline), weeks 11 and 12 (14 days), weeks 23 and 24 (14 days)
Population: Number analyzed at different time points reflects attrition due to device failure, COVID-19 restrictions, and 2 participants who withdrew after baseline
Measure: Mean (Standard Deviation); unit: % Time in Range
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 88 | 87
% Time in Range
  Baseline | 76.0 (19.2) | 72.3 (20.9)
  Week 11-12: number analyzed (Participants) | 84 | 86
  Week 11-12 | 75.2 (22.6) | 66.9 (26.2)
  Week 23-24: number analyzed (Participants) | 87 | 83
  Week 23-24 | 72.8 (23.2) | 64.7 (26.5)

3. Secondary Outcome: Glycemic Variability
Description: Glycemic variability is collected by a masked Continuous Glucose Monitor (CGM), which measures individual glucose levels every 15 minutes for two weeks via a sensor placed on the participants upper arm (underside). Glycemic variability is defined as the Standard Deviation (SD) of the mean glucose during the wear period. The range of CGM data for inclusion in this study will be 5 to 14 days, consistent with manufacturer's recommendations.
Time Frame: All 14 day periods: Run-in (2-weeks, usual-baseline), weeks 11 and 12 (14 days), weeks 23 and 24 (14 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD of mean glucose (mg/dl)
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 88 | 87
SD of mean glucose (mg/dl)
  Baseline | 39.6 (14.7) | 42.0 (13.1)
  Weeks 11-12: number analyzed (Participants) | 84 | 86
  Weeks 11-12 | 40.0 (12.9) | 44.9 (15.4)
  Weeks 23-24: number analyzed (Participants) | 87 | 83
  Weeks 23-24 | 40.8 (14.9) | 45.8 (16.3)

4. Secondary Outcome: Mean Glucose (mg/dl)
Description: A measure of the mean, 24 hour glucose concentration calculated across all recorded glucose readings during the wear period
Time Frame: All 14 day periods: Run-in (2-weeks, usual-baseline), weeks 11 and 12 (14 days), weeks 23 and 24 (14 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 88 | 87
mg/dl
  Baseline | 147.3 (42.1) | 151.4 (33.1)
  Weeks 11-12: number analyzed (Participants) | 84 | 86
  Weeks 11-12 | 149.4 (46.4) | 161.2 (50.5)
  Weeks 23-24: number analyzed (Participants) | 87 | 83
  Weeks 23-24 | 153.1 (50.7) | 162.3 (47.3)

5. Secondary Outcome: Fasting Glucose
Description: Standard (mg/dl) measure taken fasting (morning) during baseline, 12 weeks, 24 weeks
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: Number analyzed at different time points reflects attrition due to invalid lab sample, COVID-19 restrictions, and 2 participants who withdrew after baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 90 | 88
mg/dl
  Baseline | 147.5 (40.0) | 147.6 (36.2)
  Week 12: number analyzed (Participants) | 85 | 83
  Week 12 | 146.2 (41.8) | 149.3 (44.2)
  Week 24: number analyzed (Participants) | 90 | 87
  Week 24 | 149.2 (44.0) | 153.7 (51.3)

6. Secondary Outcome: Fasting Insulin (Pmol/L)
Description: Standard lab measurement for fasting insulin assessment
Time Frame: Time 0 (directly after 2-week run-in), week 12, week 24
Population: Number analyzed at different time points reflects attrition due to invalid samples, COVID-19 restrictions, and 2 participants who withdrew after baseline
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 89 | 88
pmol/L
  Baseline | 128.0 (97.1) | 138.5 (134.1)
  Week 12: number analyzed (Participants) | 84 | 81
  Week 12 | 135.7 (141.0) | 134.2 (145.0)
  Week 24: number analyzed (Participants) | 89 | 86
  Week 24 | 143.5 (145.4) | 144.2 (144.0)

7. Secondary Outcome: Fructosamine
Description: Fructosamine (umol/L) represents usual glycemia over the past 2-3 weeks, and is considered a valid marker of short term clinical glycemic patterns by the American Diabetes Association
Time Frame: Time 0 (directly after 2-week run-in),12, 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 90 | 88
umol/L
  Baseline | 273.2 (44.8) | 285.5 (42.4)
  Week 12: number analyzed (Participants) | 85 | 82
  Week 12 | 272.1 (43.5) | 286.6 (47.2)
  Week 24 | 273.0 (51.3) | 291.6 (45.8)

8. Secondary Outcome: Weight (kg)
Description: Weight measured on standardized scale in gown
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: Number analyzed at different time points 2 participants who withdrew after baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
kg
  Baseline | 102.1 (21.1) | 96.1 (21.5)
  Week 12: number analyzed (Participants) | 91 | 88
  Week 12 | 101.5 (20.4) | 95.8 (21.8)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 101.2 (20.6) | 95.9 (21.9)

9. Secondary Outcome: Total Cholesterol (mg/dL)
Description: Total cholesterol was measured as part of a lipid panel, a standard measurement for assessing clinical CVD risk
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 90 | 88
mg/dl
  Baseline | 165.9 (41.3) | 163.6 (40.9)
  Week 12: number analyzed (Participants) | 85 | 84
  Week 12 | 164.8 (39.5) | 163.6 (40.3)
  Week 24: number analyzed (Participants) | 90 | 87
  Week 24 | 161.1 (36.4) | 163.4 (40.1)

10. Secondary Outcome: Kidney Function
Description: eGFR-Cystatin-C (estimated glomerular filtration rate) = mL/min/1.73 m^2
Time Frame: Time 0 (directly after 2-week run-in),12, 24 weeks
Measure: Mean (Standard Deviation); unit: eGFR-Cystatin-C (mL/min/1.73 m^2)
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
eGFR-Cystatin-C (mL/min/1.73 m^2)
  Baseline | 83.2 (21.1) | 81.5 (20.0)
  Week 12 | 82.8 (20.5) | 80.8 (19.5)
  Week 24 | 82.0 (20.7) | 80.9 (20.7)

11. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (mmHg)
Time Frame: Time 0 (directly after 2-week run-in),12, 24 weeks
Population: Number analyzed at different time points reflects attrition due to data collection, COVID-19 restrictions, and 2 participants who withdrew after baseline
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
mmHG
  Baseline | 136.3 (15.0) | 131.9 (15.0)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 135.5 (14.8) | 129.5 (13.1)
  Week 24: number analyzed (Participants) | 84 | 83
  Week 24 | 135.6 (15.6) | 129.6 (14.8)

12. Secondary Outcome: Diastolic Blood Pressure
Description: Standard part of blood pressure measurement (mmHG)
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 89
mmHG
  Baseline | 78.5 (7.7) | 76.6 (7.4)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 78.3 (8.4) | 75.4 (7.6)
  Week 24: number analyzed (Participants) | 84 | 83
  Week 24 | 77.7 (8.6) | 75.6 (7.2)

13. Secondary Outcome: Apolipoprotein-AI
Description: Apo-AI the major protein component of high density lipoprotein (HDL)
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
mg/dL
  Baseline | 146.6 (24.3) | 150.3 (23.3)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 148.0 (25.5) | 151.0 (23.7)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 147.2 (22.5) | 152.7 (24.2)

14. Secondary Outcome: Apolipoprotein B
Description: ApoB levels indicate the atherogenic particle concentration independent of the particle cholesterol content
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
mg/dL
  Baseline | 88.0 (21.1) | 85.0 (24.0)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 88.0 (23.1) | 86.6 (25.1)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 85.4 (21.3) | 86.8 (25.8)

15. Secondary Outcome: Fibrinogen (mg/dL)
Description: A protein involved in forming blood clots in the body
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
mg/dL
  Baseline | 265.0 (51.9) | 269.3 (55.1)
  Week 12: number analyzed (Participants) | 85 | 85
  Week 12 | 268.7 (55.7) | 263.1 (50.9)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 270.4 (53.3) | 265.4 (43.2)

16. Secondary Outcome: C-reactive Protein
Description: biomarker of inflammation
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: Number of measurements over time reflect ability to collect data during covid-19 epidemic, participant dropout, and removing 3 outliers (CRP>30)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
mg/L
  Baseline | 3.93 (3.73) | 3.54 (3.27)
  Week 12: number analyzed (Participants) | 85 | 83
  Week 12 | 3.60 (3.81) | 3.56 (3.12)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 3.85 (4.42) | 3.53 (3.35)

17. Secondary Outcome: Aspartate Aminotransferase (AST) (U/L)
Description: AST (aspartate aminotransferase) is an enzyme that reflects liver function
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
U/L
  Baseline | 21.9 (9.5) | 24.9 (15.2)
  Week 12: number analyzed (Participants) | 85 | 84
  Week 12 | 22.5 (11.3) | 23.9 (15.4)
  Week 24: number analyzed (Participants) | 91 | 87
  Week 24 | 21.9 (8.7) | 23.9 (13.0)

18. Secondary Outcome: Aminotransferase (ALT) (U/L)
Description: ALT (alanine transaminase) is an enzyme, a protein that reflects liver function
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
U/L
  Baseline | 26.6 (14.5) | 28.2 (21.6)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 26.8 (15.8) | 27.1 (23.2)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 26.6 (15.0) | 26.3 (19.0)

19. Secondary Outcome: Alkaline Phosphatase (ALKPhos ) (U/L)
Description: ALP is an enzyme, a protein, that reflects liver function
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 90
U/L
  Baseline | 88.0 (41.8) | 83.3 (24.7)
  Week 12: number analyzed (Participants) | 86 | 85
  Week 12 | 90.1 (42.9) | 82.6 (24.5)
  Week 24: number analyzed (Participants) | 91 | 88
  Week 24 | 88.7 (41.9) | 83.4 (24.6)

20. Secondary Outcome: Thyroid Stimulating Hormone (TSH)
Description: Hormone measured in the blood with energy balance related role
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 90 | 87
µU/mL
  Baseline | 2.45 (1.58) | 2.17 (1.34)
  Week 12: number analyzed (Participants) | 85 | 83
  Week 12 | 2.65 (3.32) | 2.32 (1.91)
  Week 24 | 2.36 (1.66) | 2.27 (1.47)

21. Secondary Outcome: Dietary Quality (Healthy Eating Index -HEI)
Description: The Healthy Eating Index (HEI) is a measure of diet quality used to assess how well a set of foods aligns with key recommendations and dietary patterns published in the Dietary Guidelines for Americans (Dietary Guidelines). The overall HEI scores are made up of 13 components that reflect the different food groups and key recommendations in the Dietary Guidelines for Americans. The HEI is scored 0-100 (low to high), with higher scores representing greater reported intake of an overall dietary pattern aligning with USDA Dietary Guidelines. In the SODAS study, dietary intake was assessed by multiple unannounced 24-hour dietary recalls that occurred during the 2-week run-in period to assess usual habits (2 recalls over 2 weeks) and the active intervention (5 recalls over 24 weeks: 2 to 3 recalls during weeks 1-12 (period 1), and 2 to 3 recalls during weeks 13-24 (period 2). to measure any changes in diet quality. Scores during each period represent the average score of recalls.
Time Frame: Run-in period (2 weeks) - baseline, Week 1-12 (period 1), Week 13-24 (period 2).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 91 | 89
units on a scale
  Baseline | 54.7 (12.0) | 53.7 (13.6)
  Period 1: number analyzed (Participants) | 90 | 88
  Period 1 | 54.8 (13.2) | 53.1 (12.7)
  Period 2: number analyzed (Participants) | 88 | 87
  Period 2 | 53.3 (12.3) | 51.7 (13.4)

22. Secondary Outcome: The Diabetes Health Profile (DHP-18)
Description: The Diabetes Health Profile (DHP-18) is used to assess health related quality of life in diabetes across three domains (psychological distress, barriers to activity and disinhibited eating). Each item is scored on a 4-point scale, and the subscale scores are then rescaled to a 0-100 range, with higher scores indicating poorer well-being.
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 78 | 85
units on a scale
  Baseline | 79.6 (11.1) | 77.9 (11.1)
  Week 12 | 79.8 (9.98) | 78.1 (10.9)
  Week 24 | 80.6 (11.1) | 78.6 (11.7)

23. Secondary Outcome: Food Craving Inventory (FCI)
Description: The FCI is a valid and reliable self-report measure of specific food cravings. The inventory consists of 4 factors or subscales measuring cravings for high fats (8 items), carbohydrates/starches (8 items), sweets (8 items), and fast food fats (4 items), and a total score is calculated by summing the subscales. Participants rate each food on a 5-point Likert scale ranging from 0 (never) to 4 (always/almost every day). We calculated the total score by summing the individual item responses in each subscale. Higher scores indicate more frequent cravings of the 28 items.
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 78 | 80
units on a scale
  Baseline | 33.9 (15.1) | 35.4 (14.8)
  Week 12: number analyzed (Participants) | 76 | 77
  Week 12 | 29.8 (15.8) | 30.9 (15.4)
  Week 24: number analyzed (Participants) | 76 | 74
  Week 24 | 27.1 (15.9) | 31.2 (14.3)

24. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a one-month time interval. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Time Frame: Time 0 (directly after 2-week run-in), 12, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 66 | 64
units on a scale
  Baseline | 6.0 (2.7) | 6.8 (3.0)
  Week 12: number analyzed (Participants) | 66 | 60
  Week 12 | 6.0 (3.1) | 6.5 (3.1)
  Week 24: number analyzed (Participants) | 63 | 54
  Week 24 | 5.9 (2.9) | 7.1 (3.2)

25. Secondary Outcome: Medication Effect Score (MES)
Description: The medication effect score (MES) is a measure of overall diabetes regimen intensity, and is based on the dosages of medications used and their potencies. The MES is calculated for each diabetes medication in a regimen using the following equation: (actual drug dose/maximum drug dose) × drug-specific adjustment factor. The adjustment factor equates to the expected decrease in HbA1c achieved by the drug as monotherapy. The MES presumes a linear relationship between medication dosage and HbA1c, and the sum of MES values attributed to individual medications represents the maximum A1c reduction that may be expected by the regimen. It is a continuous variable with range 0 (no medications), and the maximum achievable MES is patient specific and dependent on the total number of and dose of medications reported.
Time Frame: Time 0 (directly after 2-week run-in), 6, 12, 18, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 89 | 84
units on a scale
  Week 0 | 1.64 (1.05) | 2.09 (1.40)
  Week 6: number analyzed (Participants) | 89 | 83
  Week 6 | 1.64 (1.06) | 2.05 (1.36)
  Week 12: number analyzed (Participants) | 89 | 83
  Week 12 | 1.63 (1.05) | 2.03 (1.33)
  Week 18: number analyzed (Participants) | 89 | 82
  Week 18 | 1.64 (1.06) | 2.02 (1.35)
  Week 24: number analyzed (Participants) | 87 | 82
  Week 24 | 1.64 (1.06) | 2.01 (1.36)

26. Secondary Outcome: Therapeutic Intensity Score (TIS)
Description: The therapeutic intensity score (TIS) is a summary measure that accounts for the number of medications and the relative doses a patient received to lower blood pressure. It is a continuous variable with range 0 (no medications), and the maximum achievable TIS is patient specific and dependent on the total number of antihypertensive medications reported.
Time Frame: Time 0 (directly after 2-week run-in), 6, 12, 18, 24 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diet Beverage | Water
Number analyzed (Participants) | 86 | 84
score on a scale
  Week 0 | 0.41 (0.51) | 0.42 (0.43)
  Week 6 | 0.40 (0.46) | 0.41 (0.43)
  Week 12 | 0.42 (0.49) | 0.42 (0.44)
  Week 18 | 0.41 (0.49) | 0.43 (0.45)
  Week 24 | 0.41 (0.49) | 0.42 (0.45)

ADVERSE EVENTS:
Time Frame: 26 weeks (2 week run-in period and 24-week randomized intervention period)
Arm/Group | Diet Beverage | Water
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03944616/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03944616/SAP_000.pdf